CLINICAL TRIAL: NCT04939948
Title: Multi-factor Analysis of Psychological Disorders in Patients With Inflammatory Bowel Disease
Brief Title: Multi-factor Analysis of Psychological Disorders in IBD Patients
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0332
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2021-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: inflammatory bowel disease; psychological disorders
MeSH Terms: conditions — Inflammatory Bowel Diseases; Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: None Retained — not needed

SUMMARY:
Inflammatory bowel disease IBD, including Crohn's disease (CD) and ulcerative colitis (UC), is a chronic inflammatory disease of the intestinal tract with unknown etiology. The mechanism includes environment, genetics, intestinal microecology and immunity. In recent years, the incidence of IBD in Asian countries has continued to rise, and the incidence of CD and UC in Guangzhou has reached 1.09/10 million and 2.05/10 million respectively. The patient suffers from the disease for a long time, which greatly affects the mentality and the quality of life. However, the mentality and quality of life of IBD patients have not received the attention they deserve, and research in this area is relatively lacking. The study by Lewis et al. found that among IBD patients, up to 1/3 of depression patients and 2/3 of anxiety patients were not diagnosed in time. This study conducted an Internet questionnaire survey on IBD patients diagnosed in the Department of Gastroenterology, the Second Affiliated Hospital of Zhejiang University School of Medicine, to learn about the patients 'mental and psychological state, to screen the risk factors of patients'mental and psychological diseases, and to understand the impact of mental and psychological factors on the quality of life and quality of IBD patients. The impact of the disease provides a scientific basis for the optimal treatment of IBD.

DETAILED DESCRIPTION:
Patients with IBD self-reported their disease activity using validated patient-based measures. For those with CD, the Harvey-Bradshaw Index (HBI) was utilized, and for patients with UC, the Patient-based Simple Clinical Colitis Activity Index (P-SSCAI) was employed. An HBI score greater than 4 or a P-SSCAI score of 5 or higher was classified as active disease, while an HBI score of 4 or lower or a P-SSCAI score below 5 indicated disease remission.

To assess health-related quality of life (HRQOL), participants completed the Short Health Scale (SHS), a 4-item self-management questionnaire validated for use in adult IBD patients. Each item corresponds to specific dimensions of HRQOL: symptoms, social function, disease-related worry, and general well-being. Responses were graded on a 100-mm visual analog scale, with scores ranging from 0 to 100, where higher scores represented worse HRQOL.

Participants' anxiety and depression levels were evaluated using the Generalized Anxiety Disorder-7 (GAD-7) and Patient Health Questionnaire-9 (PHQ-9)20,21. Each scale comprises 7 and 9 self-assessment items to gauge anxiety and depression, respectively. A score of GAD-7 ≥10 indicated severe anxiety symptoms, while a score of PHQ-9 ≥ 10 indicated severe depression symptoms.

The Pittsburgh Sleep Quality Index scale (PSQI) was employed to assess sleep quality, encompassing subjective sleep quality, latency, duration, efficiency, persistence, use of sleep drugs, and daytime dysfunction22. The total scores on this scale range from 0 to 21, with higher scores indicating poorer sleep quality.

Statistical analysis The survey data were collected and analyzed using IBM SPSS statistical software (version 25.0, Chicago, Illinois, USA). Quantitative data were expressed as mean and standard deviation or inter-quartile range, and group differences were compared using t-tests for normally distributed data or the Wilcoxon test for non-normally distributed data. Categorical data were presented as frequencies or percentages, and differences in frequencies between groups were assessed using the χ2 test or Fisher's exact test. The correlation between scores of GAD-7 or PHQ-9 and SHS total scores was examined using simple linear regression, and the results were presented with the coefficient R2. To study the independent effect of various variables on the quality of life (QOL), multiple regression analysis was applied. Initially, correlations between demographic and clinical variables such as age, gender, living conditions, disease status, employment, marital status, family history of IBD, GAD-7 scores, PHQ-9 scores, and SDS scores were explored using simple regression. Variables with a p-value of ≤ 0.05 in the simple regression analyses were then included in the multiple regression analysis. Odds ratios (OR), 95% confidence intervals (95% CI), and p-values were calculated for each independent variable. For all statistical tests, a two-sided p-value of 0.05 was considered the threshold for defining the level of significance.

ELIGIBILITY:
Inclusion Criteria:

Cognitive function and educational level can cooperate to complete the scale; No history of digestive system disease or mental illness;

Exclusion Criteria:

Cognitive function and educational level could not cooperate to complete the scale; Failed to fill in all the scales effectively;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were age 18 years or older, able to provide informed consent, and had sufficient knowledge to complete written questionnaires and a structured clinical interview. Participants were required to have completed their Structured Clinical Interview for Diagnostic and Statistical Manual (DSM)-IV-TR Axis I Disorders (SCID) within 4 weeks of their enrollment visit date and to meet the DSM-IV criteria for a depression or anxiety disorder.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
assess the effects of mental disease on risk of IBD-related adverse outcomes | 3 months
  assess the effects of mental disease on risk of IBD-related adverse outcomes such as IBD-related hospitalization or surgery, new or recurrent corticosteroid use, switching to an alternative anti-TNF, or death

SECONDARY OUTCOMES:
assess the effects of mental disease on drug adherence | 3 months
  assess the effects of mental disease on drug adherence such as anti-tumor necrosis factor (anti-TNF) therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Hangzhou, Zhejiang, China